CLINICAL TRIAL: NCT04584281
Title: Introduction of Artificial Intelligence (AI) and Machine Learning in Cardiotocography (CTG) Interpretation to Improve Clinical Use
Brief Title: Artificial Intelligence (AI) in Cardiotocography (CTG) Interpretation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-00501
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: To Introduce Artificial Intelligence (AI) and Machine Learning in Cardiotocography (CTG) Interpretation to Improve Clinical Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project leaders plan to create a clinical decision support (CDS) system by programming a self-learning software to analyze the cardiotocography (CTG) traces in the - already existing - database from the maternity department of the Inselspital Berne. The project leaders will process and analyze all clinical outcomes of the estimated 10000-15000 eligible patient records. CSEM will design, develop, and validate several AI architectures with the intend to create the CDS system. The AI would learn to assist on this task by training machine learning (ML) algorithms. The main purpose of the AI-CDS will be to determine the best fetal extraction moment during labor, based on a self-learning approach, as a "superhuman" support tool for obstetricians in decision making during labor.

ELIGIBILITY:
Inclusion Criteria:

* CTG-registrations of patients with singleton pregnancies during labour from 01.01.2006 to 31.12.2019
* Gestational age ≥ 24+0 weeks
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Documented refusal
* Multiple pregnancies
* CTG-registrations of planned caesarean sections

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with singleton pregnancies and CTG-registrations during labour from 01.01.2006 to 31.12.2019
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Superior prediction of fetal morbidity through the self-learning CDS system than if performed by obstetricians alone, especially in regards to specificity. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Frauenklinik Inselspital Bern, Bern, Switzerland